CLINICAL TRIAL: NCT01820325
Title: A Dose-finding Phase Ib Study Followed by a Randomized, Double-blind Phase II Study of Carboplatin and Paclitaxel With or Without Buparlisib in Patients With Previously Untreated Metastatic Non-small Cell Lung Cancer (NSCLC) of Squamous Histology
Brief Title: Safety and Efficacy of Buparlisib (BKM120) in Patients With Untreated Squamous Non-small Cell Lung Cancer
Acronym: BASALT-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to DLTs/AEs safety profile considered challenging.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBKM120D2204; 2012-005541-21 (EudraCT Number)
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Non-Small Cell Lunch Cancer
Keywords: Squamous non-small cell lung cancer; NSCLC; stage IV; BKM120
MeSH Terms: interventions — NVP-BKM120; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buparlisib + Carboplatin + Paclitaxel (Experimental): Carboplatin and paclitaxel plus buparlisib for up to 6 cycles, followed by blinded buparlisib maintenance
  Interventions: Drug: Buparlisib; Drug: Carboplatin; Drug: Paclitaxel
- Placebo + Carboplatin + Paclitaxel (Placebo Comparator): Carboplatin and paclitaxel plus buparlisib-matching placebo for up to 6 cycles, followed by blinded placebo maintenance
  Interventions: Drug: Buparlisib placebo; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Buparlisib
  Other Names: BKM120
  Arms: Buparlisib + Carboplatin + Paclitaxel
Drug: Buparlisib placebo — Placebo + Carboplatin + Paclitaxel
  Arms: Placebo + Carboplatin + Paclitaxel
Drug: Carboplatin
Drug: Paclitaxel

SUMMARY:
The Phase Ib part of the study aimed to determine the maximum tolerated dose/recommended Phase II dose (MTD/RP2D) of once daily buparlisib in combination with every-three-week carboplatin and paclitaxel in patients with previously untreated metastatic squamous NSCLC.

The purpose of the Phase II portion of the study was to assess the treatment effect of adding buparlisib versus buparlisib-matching placebo to every-three-week carboplatin and paclitaxel on progression free survival (PFS) in patients with previously untreated metastatic squamous NSCLC.

DETAILED DESCRIPTION:
Based on the observation of DLTs and AEs, the safety profile of this investigational treatment was considered challenging requiring dose reductions/interruptions and even the evaluation of an alternative schedule of buparlisib administration. The study was early terminated, and the primary objective was not met. Therefore the phase ll portion of the study was never initiated.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically and/or cytologically confirmed diagnosis of squamous NSCLC. Diagnosis of mixed squamous with a squamous component will be acceptable for enrollment.
* Patient has archival or new tumor tissue for the analysis of PI3K biomarkers
* Tumor is Stage IV at the time of signed informed consent (UICC/AJCC version 7)
* Patient has measurable or non-measurable disease according to RECIST v1.1 criteria

  • For the Phase II portion, the patient must have measurable disease according to RECIST 1.1 criteria
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 that the investigator believes is stable at the time of screening
* Patient has adequate bone marrow and organ function

Exclusion Criteria:

* Patient has received any prior systemic therapies for metastatic NSCLC. Study treatment in this clinical trial must be the patient's first systemic treatment for metastatic NSCLC. Patients are eligible if they received neo-adjuvant or adjuvant systemic therapy followed by a disease-free interval exceeding 12 months.
* Patient has symptomatic CNS metastases

  • Patients with asymptomatic CNS metastases may participate in this trial. The patient must have completed any prior local treatment for CNS metastases ≥ 28 days prior to the start of study treatment (including radiotherapy and/or surgery, or ≥14 days for stereotactic radiosurgery).
* Patient is currently receiving warfarin or other coumadin derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed.
* Patient is currently receiving treatment with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment is initiated. Switching to a different medication prior to randomization is allowed.
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others) or patients with active severe personality disorders (defined according to DSM- IV) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug
* Patient has ≥ CTCAE grade 3 anxiety
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
* Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2014-06-18 (Actual); Study Completion 2014-06-18 (Actual)

PRIMARY OUTCOMES:
Number of Total Dose-limiting Toxicity (DLT) During Dose Escalation to Determine Maximum Tolerated Dose (MTD) | Cycle 1 (21 days)
  Determine the MTD and/or RP2D of daily buparlisib in combination with paclitaxel and carboplatin in patients with advanced or metastatic squamous NSCLC.
Progression Free Survival (PFS) as measured using RECIST 1.1 | Randomization, every 6 weeks to the date of first document progression for up to 3 years
  Progression-free survival is defined as the time from randomization to the date of the first documented progression or death from any cause. The Kaplan-Meier estimate of the PFS survival function was contructed.

SECONDARY OUTCOMES:
Number of Participants With Best Overall Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors (RECIST) | Every 6 weeks from randomization until first documented progression for up to 3 years
  Overall response is the number of participants who had a complete response (CR) or a partial response (PR) based on local investigator's assessment of RECIST criteria. Per RECIST: CR, all detectable tumor has disappeared; PR, a >=30% decrease in the sum of the longest dimensions of the target lesions (TLs) taking as a reference the baseline sum, no worsening of non-TLs, and no new lesions; Progressive disease (PD), a >=20% increase in TLs, clearly worsening of non-TLs, or emergence of new lesions; Stable Disease (SD), small changes that do not meet previously given criteria.
Overall Survival Time | Every 6 weeks from randomization until first documented progression for up to 3 years
  Overall survival (OS) time was measured from the start of study drug to the date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last contact. Data was collected post treatment every 6 weeks until approximately 75% of patients have reached the survival endpoint (Phase I + Phase II).
Time to overall response | Every 6 weeks from randomization until first documented progression for up to 3 years
  Time to overall response (TTR) is defined as the time from the date of first drug intake in Phase Ib and from the date of randomization in Phase II to the date of first documented response. TTR will primarily be listed.
The Overall Safety and Tolerability of buparlisib (BKM120) | Screening, Until 30 days after last dose
  Assessments consisted of recording all AEs and serious adverse events (SAEs), the regular monitoring of hematology, blood chemistry, vital signs, physical condition and body weight.
Change From Baseline in Quality of Life Measured by the Functional Assessment of EORTC QLQ- C-30 and lung cancer module (QLQ-LC-13) | Screening, Every 6 weeks until disease progression for up to 3 years
  Quality of life (QoL) is evaluated using EORTC QLQ-C30 and QLQ-LC-13 scale. QLQ-L30 is composed of 30 items, whose responses range from 0 to 4. The QLQ-LC13 is used in conjucntion with the QLQ-C30 and provides information on an additional 13 items specifically relating to lung cancer. It incorporates one multi-item scale to assess dyspnea and a series of single-item scale to assess pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and haemoptysis. All the multi-item scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Time to deterioration by the Functional Assessment of EORTC QLQ- C-30 and lung cancer module (QLQ-LC-13) | Screening, Every 6 weeks until disease progression for up to 3 years
  Time to definitive 10% deterioration in the global health status / QoL, physical functioning, emotional functioning, social functioning, and lung cancer symptoms scales will be assessed in the two treatment arms.
Buparlisib concentrations | Cycle 1 day 8 and 15, Cycle 2 day 1, Cycle 7-Cycle n, day 1
  Pharmacokinetics of buparlisib will be investigated in order to investigate any unexpected impact of carboplatin and paclitaxel therapy on the pharmacokinetics of buparlisib. For this purpose, plasma samples will be collected during phase II of the trial. In one set of the population (N=40) samples will be collected according to a sparse sampling strategy over the entire course of the treatment, to allow a proper estimate of the pharmacokinetic parameters. In addition, trough samples should be collected, for the whole population, for measurement of buparlisib/placebo. These additional samples will allow investigating potential PK/PD relationships for various therapeutic or adverse outcome in the whole study population.
Duration of overall response | Every 6 weeks from randomization until first documented progression for up to 3 years
  Duration of overall response (DR) is defined as the elapsed time between the date of first documented response and the following date of event defined as the first documented progression or death due to underlying cancer. DR will primarily be listed. DR may be described using Kaplan-Meier curves and any related statistics if relevant and will be presented by treatment group in phase II. These analyses will be performed on the responder subset, i.e. patients with a confirmed complete response (CR) or partial response (PR).
Characterize the PK of buparlisib under alternative dosing regimen when combined with paclitaxel and carboplatin in the target population | cycle 1 to 6 in Phase Ib portion
  Buparlisib concentrations and model-based PK derived parameters

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (2):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Northwest Cancer Specialists Compass Oncology -BKM, Portland, Oregon
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Ulm, Germany
- Novartis Investigative Site, Napoli, Italy
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

REFERENCES:
- [Derived] Vansteenkiste JF, Canon JL, De Braud F, Grossi F, De Pas T, Gray JE, Su WC, Felip E, Yoshioka H, Gridelli C, Dy GK, Thongprasert S, Reck M, Aimone P, Vidam GA, Roussou P, Wang YA, Di Tomaso E, Soria JC. Safety and Efficacy of Buparlisib (BKM120) in Patients with PI3K Pathway-Activated Non-Small Cell Lung Cancer: Results from the Phase II BASALT-1 Study. J Thorac Oncol. 2015 Sep;10(9):1319-1327. doi: 10.1097/JTO.0000000000000607. PMID 26098748